CLINICAL TRIAL: NCT00006367
Title: Autologous Peripheral Blood Stem Cell Mobilization and Transplantation for Myelofibrosis
Brief Title: Chemotherapy Followed by Peripheral Stem Cell Transplantation in Treating Patients With Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1006.00; FHCRC-1006.00; MCC-12245; MCC-IRB-5698; NCI-G00-1866; CDR0000068240 (Registry Identifier: PDQ)
Record Dates: First submitted 2000-10-04; First posted 2003-11-11 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2010-06

CONDITIONS: Chronic Myeloproliferative Disorders
Keywords: polycythemia vera; chronic idiopathic myelofibrosis; essential thrombocythemia
MeSH Terms: conditions — Myeloproliferative Disorders; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential | interventions — Filgrastim; Busulfan; Cytarabine; Idarubicin; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: busulfan
Drug: cytarabine
Drug: idarubicin
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy followed by peripheral stem cell transplantation in treating patients who have myelofibrosis.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the ability of myeloablative chemotherapy followed by peripheral blood stem cell (PBSC) transplantation to restore effective marrow hematopoieses in patients with advanced idiopathic myelofibrosis or myelofibrosis secondary to other myeloproliferative disorders. II. Determine the ability of this regimen to palliate symptoms and prolong survival in these patients. III. Determine if there is evidence of clonal hematopoieses before PBSC mobilization, in the PBSC product, and after transplantation in these patients. IV. Correlate the properties of the peripheral blood before mobilization and the PBSC product with engraftment in these patients. V. Correlate the markers of angiogenesis with clinical parameters in these patients.

OUTLINE: Patients with evidence of leukemic progression receive cytoreduction therapy consisting of idarubicin IV on days 1-3 and cytarabine IV continuously over days 1-7 followed by filgrastim (G-CSF) subcutaneously (SC) daily until blood counts recover and leukapheresis is completed. Patients undergo leukapheresis beginning when blood counts recover and continuing until the target number of cells are collected. Patients with no evidence of leukemic progression receive filgrastim SC daily until leukapheresis is completed. Patients undergo leukapheresis beginning on day 4 and continuing until the target number of cells are collected. Patients receive myeloablative therapy consisting of oral busulfan every six hours on days -5 to -2. Patients with leukemic progression begin myeloablative therapy at least 28 days after completion of chemotherapy. Patients receive autologous peripheral blood stem cells IV on day 0. Patients are followed at 1 month, 3 months, 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 10-44 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of idiopathic myelofibrosis or other myeloproliferative disorder with myelofibrosis Evidence of advanced disease or hematologic abnormalities due to severe fibrosis such as 1 or more of the following poor prognostic factors: Hemoglobin less than 10 g/dL Platelet count less than 100,000/mm3 WBC less than 4,000/mm3 Symptomatic splenomegaly Constitutional symptoms inadequately controlled with low dose chemotherapy Abnormal karyotype Patients without evidence of advanced disease undergo PBSC harvest and transplantation is delayed until there is evidence of disease progression Leukemia progression (greater than 15% peripheral blood blasts) allowed if the history of a chronic myeloproliferative disorder of at least 6 months duration is well documented Ineligible for or refusal of allogeneic transplantation No other cause of myelofibrosis other than myeloproliferative disorders, such as the following: Metastatic carcinoma Lymphoma Hairy cell leukemia Myelodysplastic syndrome De novo acute leukemia Collagen vascular disorders Granulomatous infections

PATIENT CHARACTERISTICS: Age: 75 and under Performance status: Not specified Life expectancy: Not specified Hematopoietic: See Disease Characteristics WBC no greater than 30,000/mm3 (may be reduced to less than 30,000/mm3 using hydroxyurea or induction chemotherapy) Hepatic: Bilirubin no greater than 2 times upper limit of normal (ULN)* Transaminases no greater than 2 times ULN* * Unless due to extramedullary hematopoiesis in the liver Renal: Creatinine no greater than 2 times normal OR Creatinine clearance at least 50% Cardiovascular: No prior or active congestive heart failure* LVEF at least 50%* *If receiving study cytoreductive therapy Pulmonary: Total lung capacity at least 50% predicted OR Corrected DLCO at least 50% predicted Other: No active infection No poorly controlled seizure disorders Not pregnant or nursing Negative pregnancy test Fertile patients must use effective barrier contraception HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: See Disease Characteristics At least 7 days since prior hydroxyurea Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-05; Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne E. Anderson, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (9):
- United States (7):
  - Katmai Oncology Group, Anchorage, Alaska
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of Illinois College of Medicine, Chicago, Illinois
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Washington University Siteman Cancer Center, St Louis, Missouri
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Hopital Saint-Louis, Paris, France
- Addenbrooke's NHS Trust, Cambridge, England, United Kingdom

REFERENCES:
- [Result] Anderson JE, Tefferi A, Craig F, Holmberg L, Chauncey T, Appelbaum FR, Guardiola P, Callander N, Freytes C, Gazitt Y, Razvillas B, Deeg HJ. Myeloablation and autologous peripheral blood stem cell rescue results in hematologic and clinical responses in patients with myeloid metaplasia with myelofibrosis. Blood. 2001 Aug 1;98(3):586-93. doi: 10.1182/blood.v98.3.586. PMID 11468154